CLINICAL TRIAL: NCT00141193
Title: Clinical Protocol For a Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Celecoxib (SC-58635) In The Prevention of Colorectal Sporadic Adenomatous Polyps (PRESAP)
Brief Title: Prevention of Colorectal Sporadic Adenomatous Polyps (PRESAP)
Acronym: PRESAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EQ4-00-02-018; A3191107
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Colorectal Adenoma
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Placebo Comparator)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
This study is a prospective, randomized, double-blind, placebo-controlled, multi-center trial to compare the efficacy and safety of celecoxib 400mg QD versus placebo in reducing the occurrence of new colorectal adenomas post-polypectomy at Month 13 (Year 1) and Month 37 (Year 3) of study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* The subject has had a documented colonoscopy to the cecum performed by a study-related physician with adequate preparation resulting in diagnosis and clearance of an adenomatous polyp(s) within 4 months prior to randomization.
* The subject is willing to abstain from chronic use of all NSAIDs or COX-2 inhibitors excluding aspirin at cardioprotective doses for the duration of the study.

Exclusion Criteria:

* The subject has a history of Familial Adenomatous Polyposis or Hereditary Non-Polyposis Colorectal Cancer.
* The subject has a history of inflammatory bowel disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1561 (Actual)
Dates: Start 2001-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of celecoxib in reducing the proportion of subjects with new colorectal adenomas post baseline polypectomy after Month 13 (Year 1) and Month 37 (Year 3) of study drug administration. | 3 years

SECONDARY OUTCOMES:
The number of colorectal adenomas in study subjects | 3 years
the histopathologic grade of colorectal adenomas | 3 years
the size of colorectal adenomas measured after one year and three years of study drug use. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (8):
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Kiego, California
  - Pfizer Investigational Site, North Chicago, Illinois
  - Pfizer Investigational Site, Oak Park, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Richmond, Virginia
- Australia (2):
  - Pfizer Investigational Site, Townsville, Queensland
  - Pfizer Investigational Site, Geelong, Victoria
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (6):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Abbotsford, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, St. John's
- Pfizer Investigational Site, Santiago, RM, Chile
- Pfizer Investigational Site, Beijing, China
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Liberec
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Arhus C, Denmark
- Pfizer Investigational Site, Oulu, Finland
- France (4):
  - Pfizer Investigational Site, Bobigny
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
- Germany (9):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Freising
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Künzing
  - Pfizer Investigational Site, Ludwigshafen
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Ulm
- Hong Kong (2):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, New Territories
- Hungary (2):
  - Pfizer Investigational Site, Győr
  - Pfizer Investigational Site, Szekszárd
- Ireland (2):
  - Pfizer Investigational Site, Wilton, Cork
  - Pfizer Investigational Site, Dublin
- Israel (8):
  - Pfizer Investigational Site, Beer-Sheeva
  - Pfizer Investigational Site, Hadera
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Hashomer
  - Pfizer Investigational Site, Holon
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Aviv
- Italy (5):
  - Pfizer Investigational Site, San Giovanni Rotondo, Italy/Foggia/Italy
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Siena
- Pfizer Investigational Site, Maastricht, Netherlands
- Pfizer Investigational Site, Skien, Norway
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Pfizer Investigational Site, Warsaw, Poland
- Pfizer Investigational Site, Lisbon, Portugal
- Pfizer Investigational Site, Moscow, Russia
- Pfizer Investigational Site, Singapore, Singapore
- Pfizer Investigational Site, Bratislava, Slovakia
- South Africa (2):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Cape Town, Western
- Spain (5):
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Donostia / San Sebastian, Guipuzcoa
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Seville, Sevilla
- Sweden (2):
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- Pfizer Investigational Site, Geneva, Switzerland
- Pfizer Investigational Site, Kaohsiung City, Taiwan
- United Kingdom (4):
  - Pfizer Investigational Site, Newport, Gwent
  - Pfizer Investigational Site, Harrow, Middlesex
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Oxford
- Pfizer Investigational Site, Montevideo, Uruguay

REFERENCES:
- [Derived] Arber N, Lieberman D, Wang TC, Zhang R, Sands GH, Bertagnolli MM, Hawk ET, Eagle C, Coindreau J, Zauber A, Lanas A, Levin B. The APC and PreSAP trials: a post hoc noninferiority analysis using a comprehensive new measure for gastrointestinal tract injury in 2 randomized, double-blind studies comparing celecoxib and placebo. Clin Ther. 2012 Mar;34(3):569-79. doi: 10.1016/j.clinthera.2012.02.001. Epub 2012 Mar 2. PMID 22386831
- [Derived] Arber N, Spicak J, Racz I, Zavoral M, Breazna A, Gerletti P, Lechuga MJ, Collins N, Rosenstein RB, Eagle CJ, Levin B. Five-year analysis of the prevention of colorectal sporadic adenomatous polyps trial. Am J Gastroenterol. 2011 Jun;106(6):1135-46. doi: 10.1038/ajg.2011.116. Epub 2011 Apr 19. PMID 21503000
- [Derived] Solomon SD, Wittes J, Finn PV, Fowler R, Viner J, Bertagnolli MM, Arber N, Levin B, Meinert CL, Martin B, Pater JL, Goss PE, Lance P, Obara S, Chew EY, Kim J, Arndt G, Hawk E; Cross Trial Safety Assessment Group. Cardiovascular risk of celecoxib in 6 randomized placebo-controlled trials: the cross trial safety analysis. Circulation. 2008 Apr 22;117(16):2104-13. doi: 10.1161/CIRCULATIONAHA.108.764530. Epub 2008 Mar 31. PMID 18378608
- [Derived] Arber N, Eagle CJ, Spicak J, Racz I, Dite P, Hajer J, Zavoral M, Lechuga MJ, Gerletti P, Tang J, Rosenstein RB, Macdonald K, Bhadra P, Fowler R, Wittes J, Zauber AG, Solomon SD, Levin B; PreSAP Trial Investigators. Celecoxib for the prevention of colorectal adenomatous polyps. N Engl J Med. 2006 Aug 31;355(9):885-95. doi: 10.1056/NEJMoa061652. PMID 16943401
- [Derived] Solomon SD, Pfeffer MA, McMurray JJ, Fowler R, Finn P, Levin B, Eagle C, Hawk E, Lechuga M, Zauber AG, Bertagnolli MM, Arber N, Wittes J; APC and PreSAP Trial Investigators. Effect of celecoxib on cardiovascular events and blood pressure in two trials for the prevention of colorectal adenomas. Circulation. 2006 Sep 5;114(10):1028-35. doi: 10.1161/CIRCULATIONAHA.106.636746. PMID 16943394
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EQ4-00-02-018&StudyName=Prevention%20of%20Colorectal%20Sporadic%20Adenomatous%20Polyps%20%28PRESAP%29